CLINICAL TRIAL: NCT02969031
Title: Improving Communication Between Cancer Patients and Oncologists Using Patient Feedback on Actual Conversations and the ABIM Maintenance of Certification Program
Brief Title: Improving Communication Between Cancer Patients & Oncologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Board of Internal Medicine (Other); Duke University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, James A. Tulsky, Chair, Department of Psychosocial Oncology and Palliative Care, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-099
Record Dates: First submitted 2016-11-16; First posted 2016-11-21 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Cancer
Keywords: communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced SCOPE training (Experimental): Complete a baseline questionnaire, administer satisfaction surveys anonymously to a sample of their patients, audio record (using a smartphone application) eight clinic visits with eight different patients. Receive survey feedback as well as the enhanced SCOPE program that provides feedback on their audio-recorded encounters via a web-based interactive program.
  Interventions: Behavioral: Enhanced SCOPE training
- Standard Communication training (Active Comparator): Complete a baseline questionnaire, administer satisfaction surveys anonymously to a sample of their patients. Receive the results of the patient surveys and be asked to conduct a quality improvement activity of their own design that responds to the feedback (the current "standard" communication PIM).
  Interventions: Behavioral: Standard Communication training

INTERVENTIONS:
Behavioral: Enhanced SCOPE training — Intervention is integrated into the American Board of Internal Medicine (ABIM) Maintenance Of Certification (MOC) process.
  Arms: Enhanced SCOPE training
Behavioral: Standard Communication training — Standard Communication training
  Arms: Standard Communication training

SUMMARY:
The overarching goal of this project is to improve communication between oncologists and their patients by ensuring that the patient's voice is heard in the medical encounter. Thus, the hope is to improve the experience for patients living with cancer. The investigators seek to accomplish this goal by providing oncologists communication skills training that includes feedback on their own audio-recorded conversations. The feedback will come from two sources: 1) Professional research assistant coders who will identify objective learning opportunities based on specific coding criteria and 2) Trained patient reviewers who will listen to the recordings and offer their own, subjective feedback at key moments in the encounters.

DETAILED DESCRIPTION:
The primary objective of the Enhanced SCOPE program is to teach oncologists to recognize the role of emotion in discussions with cancer patients, to increase their self-efficacy for addressing affective concerns, and to provide them with the skills for doing so. Oncologists are most likely to achieve competency in these areas when, in addition to didactic training, they can also observe their own conversation and receive feedback on their interactions. The Enhanced SCOPE program itself is an online web application that can be viewed from any computer with internet connectivity. The investigators will be conducting a randomized controlled trial to test the impact on patient satisfaction and medical visit quality of a communication skills teaching intervention for oncologists that is integrated into the American Board of Internal Medicine (ABIM) Maintenance Of Certification (MOC) process. Oncologists who choose to enroll in this pilot Practice Improvement Module (PIM) will complete a baseline questionnaire, send out satisfaction surveys to a sample of their patients, and then audio record (using a smartphone application) eight clinic visits with eight different patients. Oncologists who are assigned to the control arm will receive the results of the patient surveys and be asked to conduct a quality improvement activity that responds to the feedback (the current "standard" communication PIM). Oncologists assigned to the intervention arm will receive the survey feedback as well as the enhanced SCOPE program that provides feedback on their audio-recorded encounters via a web based interactive program. The feedback will come from two sources: 1) Professional research assistant coders who will identify objective learning opportunities based on specific coding criteria (e.g., empathic opportunities, use of open-ended questions) and 2) Trained patient reviewers who will listen to the recordings and offer their own, subjective feedback at key moments in the encounters. These patient reviewers will be drawn from our stakeholder partners and are active patient advocates. They will be treated as members of the research team, paid for the reviews, and are not patients of the study physicians. One month after reviewing their feedback, oncologists in both arms will audio record another eight encounters and send out satisfaction surveys to a new sample of patients.

ELIGIBILITY:
Inclusion Criteria:

* All American Board of Internal Medicine (ABIM) Board certified oncologists practicing in the U. S. and enrolled in Maintenance of Certification.
* Have a study-compatible smart phone.
* Eligible patients will have metastatic cancer.
* At least 18 years of age.
* Speak and read English.
* Receive oncology care from an enrolled oncologist.

Exclusion Criteria:

* Dana Farber Cancer Institute oncologists and oncologists who do not speak English to their patients.
* Patients who do not speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tulsky, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Patient-Centered Outcomes Research Institute (PCORI) Research Award Listing — http://www.pcori.org/research-results/2014/improving-communication-between-cancer-patients-and-oncologists-using-patient
- See also: Dana Farber Cancer Institute (DFCI), Department of Psychosocial Oncology and Palliative Care (POPC) Listing of Current Research and PCORI Award — https://www.dana-farber.org/research/departments-centers-and-labs/departments-and-centers/department-of-psychosocial-oncology-and-palliative-care/research/
- See also: Vital Talk is a non-profit whose mission is to nurture healthier connections between patients and clinicians. We are using Vital Talk intellectual property (e.g., REMAP) for the intervention — https://www.vitaltalk.org/

RESULTS

PARTICIPANT FLOW:
Period: Enrolled and Randomized
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 73 | 75
Completed | 73 | 75
Not Completed | 0 | 0
Period: Collection of Baseline Surveys
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 73 | 75
Completed | 34 | 23
Not Completed | 39 | 52
Period: Collection of Baseline Recordings
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 34 | 23
Completed | 22 | 18
Not Completed | 12 | 5
Period: Completed Intervention
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 22 | 18
Completed | 15 | 14
Not Completed | 7 | 4
Period: Collection of Follow-Up Surveys
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 15 | 14
Completed | 15 | 12
Not Completed | 0 | 2
Period: Collection of Follow-Up Recordings
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 15 | 12
Completed | 15 | 12
Not Completed | 0 | 0
Period: Completed and Analyzed
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Started | 15 | 12
Completed | 15 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced SCOPE Training | Standard Communication Training | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.00 (9.8) | 51.92 (9.0) | 52.52 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 12 | 11 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Religion [Count of Participants; unit: Participants]
  Christian | 9 | 8 | 17
  Jewish | 0 | 1 | 1
  Islamic/Muslim | 1 | 2 | 3
  Buddhist/Hindu/Eastern | 1 | 0 | 1
  No Affiliation | 4 | 1 | 5
Previous Training [Count of Participants; unit: Participants]
  Medical School | 4 | 4 | 8
  Residency | 4 | 3 | 7
  Fellowship | 2 | 4 | 6
  Practice Training | 6 | 2 | 8
  No Previous Training | 5 | 5 | 10
Social vs. Technical Inclination [Count of Participants; unit: Participants]
  Social and Behavioral | 10 | 5 | 15
  Technical and Scientific | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Provider to Patient Communication Score
Description: The score measures the construct of patient's perception of attentive response by the medical oncologist during recalled office encounters over 12 months. Patients completed the Clinician Group Consumer Assessment of Healthcare Providers and Systems (CG-CAHPS©) Version 1.0 questionnaire via computer or phone Interactive Voice Response (IVR) system.The Provider to Patient Communication Score:(1) Provider explained things in a way that was easy to understand (2) Provider listened carefully to patient (3) Provider showed respect for what patient had to say (4) Provider spent enough time with patient. Coded as 1 (Yes, definitely), 2 (Yes, somewhat), 3 (No), or 4 (I prefer not to answer).Obtained aggregate score ((1) to (3) above), calculated avg. of the scores to each question. Avgs. modeled with linear mixed-effect model. Analyzed data in both cases where a) missing responses are dropped from data and b) missing responses are kept in dataset. Lower score indicates more desirable outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Number analyzed (Participants) | 15 | 12
score on a scale | 1.0423 (0.1380) | 1.0723 (0.2049)

2. Secondary Outcome: Empathic Response to Patient Expressions of Negative Emotions
Description: What does the outcome measure? The outcome measures the construct of a physician's skill at providing appropriate empathic responses to patient's expressions of emotional concerns. The measure is the ratio of the number of empathic responses to the total empathic opportunities that occur during a provider-patient encounter.
  How is the outcome measured? The provider-patient encounters are audio recorded. Trained listeners review, score and code the physician responses from the audio-recorded conversations. This code indicates an empathic opportunity. Behaviors that represent appropriate empathic responses are also coded.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: # empathic responses/# empathic opportun
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
Number analyzed (Participants) | 15 | 12
# empathic responses/# empathic opportun | 0.2054 (0.2678) | 0.1203 (0.2735)

ADVERSE EVENTS:
Description: The number of participants at risk for adverse events is 0 because this is a social/behavioral research trial, not a clinical trial, and therefore there is no medical risk to participants to 0 Total number of participants at risk- e.g. All-Cause Mortality, Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Enhanced SCOPE Training | Standard Communication Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT02969031/Prot_SAP_000.pdf